CLINICAL TRIAL: NCT04366570
Title: Neck-shoulder Pain - is it Possible to Use Commonly Used Provocative Tests and Functional Scores for Evaluation? Large Scale Prospective Cohort Study
Brief Title: Neck-shoulder Pain. Large Scale Prospective Cohort Study
Acronym: NSP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Lipina Marina Mikhailovna, associate professor, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 07-18
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Neck, Shoulder and Arm Syndrome
Keywords: neck, shoulder, cervical spine, sagittal balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The 1st group: (n=511; 36,45%) included patients with extra-articular injury of the proximal humerus (rotator cuff tear, anatomical and surgical neck fracture)
  Interventions: Other: clinical assessment of the shoulder and the cervical spine includes stress guideline tests
- The 2nd group: (n=309; 22,04%) included patients with intra-articular injury of the proximal humerus (contracture of the shoulder joint and shoulder instability, humeral head fracture, including Hill-Sachs lesion)
  Interventions: Other: clinical assessment of the shoulder and the cervical spine includes stress guideline tests
- The 3rd group: (n=582; 41,51%) - patients with injury of subacromial (suprahumeral) space (soft tissue injury, acromioclavicular and sternoclavicular joint injury, diaphyseal and distal end clavicle fracture)
  Interventions: Other: clinical assessment of the shoulder and the cervical spine includes stress guideline tests

INTERVENTIONS:
Other: clinical assessment of the shoulder and the cervical spine includes stress guideline tests — As a result of statistical processing, we are planning to obtain the most sensitive and specific tests from the clinical examination protocol

SUMMARY:
The aim of this study is to determine and statistically justify the correlation between shoulder girdle injuries and the development of neck-shoulder pain syndrome.

The study enrolled 1402 patients with hospital-treated shoulder girdle injuries (with consequences of upper limb trauma). Detailed protocol and questionnaire for clinical examination after discharge from the hospital were conducted. The prevalence of neck-shoulder pain among patients was calculated. The diagnostic value (sensitivity and specificity) of tests used in the study was assessed.

DETAILED DESCRIPTION:
The study's objective is to investigate and statistically justify the correlation between shoulder girdle injury (and its treatment) and NSP in patients without previous pathology.

Methods. Study design. This study was prospective, cohort, single center. A total of 1402 consecutive patients (with consequences of upper limb trauma) - 1014 males (72,3%) and 388 females (27,7%) aged 18-60 years (mean 40,5 ± 3,8 years) referred for shoulder examinations in our musculoskeletal clinic since 2013 were included.

The study was approved by the institutional Ethical Committee. Patient inclusion criteria: male and female individuals aged 18 to 60 years old; the shoulder girdle injury at least 1 year ago plus surgical or conservative injury-related treatment; patients able and willing to actively participate to the necessary rehabilitation protocol and clinical and radiological procedures; signed an ethics committee reviewed and approved informed consent form.

Patient exclusion criteria: previous spine injuries and diseases; combined distal and midshaft humerus fractures; patients unwilling to participate to the study.

Assessment methods. The patients were divided into 3 study groups according to localization of the injury.

The 1st group (n=511; 36,45%) included patients with extra-articular injury of proximal humerus (rotator cuff tear, anatomical and surgical neck fracture).

The 2nd group (n=309; 22,04%) included patients with intra-articular injury of proximal humerus (contracture of the shoulder joint and shoulder instability, humeral head fracture, including Hill-Sachs lesion) and the 3rd group (n=582; 41,51%) - patients with injury of subacromial (suprahumeral) space (soft tissue injury, acromioclavicular and sternoclavicular joint injury, diaphyseal and distal end clavicle fracture).

Totally, surgical treatment was performed in 771 cases (55%) and 631 patients (45%) were given conservative treatment. 220 patients (28,5%) in group 1, 155 patients (20,1%) in group 2 and 396 patients (51,4%) in group 3 received surgery. Likewise, 291 patients (46,1%) in group 1, 154 patients (24, 4%) in group 2 and 186 patients (29,5%) in group 3 were treated conservatively.

Since in our research we examined patients who had late posttraumatic/postoperative complications, special scales, survey questionnaires, and physical examination were conducted. Methods were performed at three points of the study: 1 year, 1,5 years and 2 years after discharge from the hospital.

On the first point (1 year after discharge) physical examination of all the patients and questionnaire assessments were performed. In some cases, the questionnaires were conducted via mobile phone with the subsequent visit for physical examination. At 6-8 months after the first visit, the next point of the research was performed. The questionnaires used in point 1 were administered. The patients who demonstrated a decrease in questionnaire scales rates were invited for clinical re-examination 1,7-2,2 years after the injury.

Pain intensity was evaluated using the following scales: VAS (visual analogue scale), UCLA (University of California Los Angeles) and SPADI (The Shoulder Pain and Disability Index).

Humeral articulation function was evaluated using following scales: UCLA (University of California Los Angeles), SPADI (The Shoulder Pain and Disability Index) and DASH (Disabilities of the Arm, Shoulder and Hand).

Shoulder function was evaluated using following scales: UCLA (University of California Los Angeles), SPADI (The Shoulder Pain and Disability Index) and DASH (Disabilities of the Arm, Shoulder and Hand).

ODI (Oswestry Disability Index) and SF-36 (Short Form-36 Health Status Survey) were used for disability and life quality assessment, respectively.

We set commonly used clinical tests to conduct the protocol for shoulder joint and cervical spine investigation. To investigate the shoulder girdle a number of tests was performed: stress test, range of motion test, test for shoulder bursitis, test for shoulder instability, test for rotator cuff injury, tests for acromioclavicular joint and long head of the biceps tendon pathology, etc. Cervical spine examination included range of motion, flexibility, pain localization and sagittal balance assessment. As a result, the protocol consisted of 15 tests for examination of the shoulder girdle and 10 tests for assessment of the cervical spine: Test (T) 1 - rotation mobility test, Т2 - test of head rotation in maximum extension, Т3 - test of head rotation in maximum flexion, Т4 - percussion test, Т5 - O'Donoghue test, Т6 - cervical spine distraction test, Т7 - shoulder press test, Т8 - test of maximum compression of the intervertebral foramina Т9 - Jackson compression test, Т10 - intervertebral foramina compression test, Т11 - quick test of combined motion, Т12 - Codman sign, Т13 - long head of the biceps tendon speed test, Т14 - Dawbarn sign, Т15 - Jobe supraspinatus test, Т16 - Gerber's lift-off test, Т17 - supine Napoleon test (belly-press test), Т18 - teres test, Т19 - nonspecific supraspinatus test, Т20 - painful arc, Т21 - Neer impingement sign, Т22 - Dugas, Т23 - O'Brien active compression test, Т24 - apprehension test, Т25 - Gerber-Ganz anterior drawer test; each test was scored.

ELIGIBILITY:
Inclusion Criteria:

male and female individuals aged 18 to 60 years old; the shoulder girdle injury at least 1 year ago plus surgical or conservative injury-related treatment; patients able and willing to actively participate to the necessary rehabilitation protocol and clinical and radiological procedures; signed an ethics committee reviewed and approved informed consent form.

Exclusion Criteria:

previous spine injuries and diseases; combined distal and midshaft humerus fractures; patients unwilling to participate to the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 1402 consecutive patients (with consequences of upper limb trauma) - 1014 males (72,3%) and 388 females (27,7%) aged 18-60 years (mean 40,5 ± 3,8 years) referred for shoulder examinations in our musculoskeletal clinic since 2013 were included.
Sampling Method: Non-Probability Sample
Enrollment: 1402 (Actual)
Dates: Start 2013-01-12 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
correlation between shoulder girdle injury (and its treatment) and NSP in patients without previous pathology | 1-2 years after injury
  To carry out these tasks, it seems important to define and statistically substantiate the connection between shoulder injuries and the development of NSP in patients without vertebrogenous pathology. Then to analyze the diagnostic value (sensitivity and specificity) of the most used and well known cervical and shoulder clinical tests and stress tests. Based on the data and the statistical distribution of results, identify the most used clinical types of NSP, and create a working classification of it.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Lychagin, MD, PhD, Study Chair — IM Sechenov University; Eugene B Kalinsky, MD, PhD, Principal Investigator — IM Sechenov University